CLINICAL TRIAL: NCT05459961
Title: Randomized, Double-Blind, Crossover Study to Assess the Effects of a Spermidine Supplement on Metabolomics in Older Men
Brief Title: Metabolic Responses to Spermidine Supplementation.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chrysea Labs Lda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIO2203
Record Dates: First submitted 2022-07-01; First posted 2022-07-15 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Spermidine

STUDY DESIGN:
Intervention Model Description: randomised double blind placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active (Active Comparator): oral spermidine supplement
  Interventions: Dietary Supplement: oral spermidine
- placebo (No Intervention): matching placebo

INTERVENTIONS:
Dietary Supplement: oral spermidine — oral supplement
  Arms: active

SUMMARY:
Spermidine is naturally present in cells, organs, circulating cardiovascular system, and as part of our normal dietary intake. Studies suggest Spermidine is involved in antioxidation, autophagy, apoptosis, and immune regulation. Spermidine is typically present in foods of plant origin, such as natto, beans, fruits, vegetables, cheese, potatoes, bread, and cereals. Adequate spermidine dietary intake is important, given evidence of declining spermidine levels with age in humans and other species, and the evidence for positive effects of spermidine supplementation on age related biology.

To date, human research studies utilised extracts containing low levels of spermidine (< 10%) and multiple other constituents, but this study will use pure spermidine to explore relevant mechanisms of action, biological effects, and identify potential biomarkers of positive biological effects.

DETAILED DESCRIPTION:
This is a placebo controlled, double blind, randomised, within subject controlled study of supplementation with oral spermidine or placebo each for up to four weeks. The primary objective of this exploratory study is to examine the safety and biological effects of this pure full-dose spermidine supplement on metabolomics, inflammatory and metabolic markers, and transcriptomics.

Study subjects are generally healthy males aged 50-70 After screening, subjects will enter a two week run-in (stabilisation) phase and then be randomised to blinded active or placebo for the first one week supplementation period. After a washout period, subjects will receive either blinded placebo or active for a second supplementation period of up to four weeks. The full study will require six visits by each study subject to the study site over a period of nine weeks, for blood and urine samples, and dietary intake assessments.

Subjects are required to maintain a normal consistent dietary intake during the study and abstain from alcohol in the 24 hours before study visits.

Assays include routine haematology and chemistry, CRP (C reactive protein), lipid screen, serum and urine metabolomics and polyamines, lipidomics, transcriptomics, and autophagy assays.

ELIGIBILITY:
Inclusion Criteria:

Caucasian men, 50-70 years of age

Non-user or former users (cessation ≥6 months) of nicotine products (e.g., cigarettes, chewing tobacco) during the study period.

Non-user or former users (cessation ≥6 months) of any marijuana or hemp products and no plans to use marijuana or hemp products during the study period

Willing to maintain physical activity and exercise patterns, body weight, and habitual diet throughout the trial.

No health conditions that would prevent the subject from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history, physical examination, and routine laboratory test results.

Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

Abnormal laboratory test results of clinical significance

Clinically important gastrointestinal (GI) condition that would potentially interfere with the evaluation of the study product

Type I or Type II diabetes mellitus.

Uncontrolled pulmonary (including uncontrolled asthma), cardiac, hepatic, renal, endocrine, hematologic, immunologic, or neurologic disease.

Had a positive SARS-CoV2 (COVID) test and experienced symptoms for > 2 months (i.e. long COVID)

Has a condition the Clinical Investigator believes would interfere with ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-08-14 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the safety and effects of a high purity Spermidine supplement in healthy older men. | Baseline, and after one, three, four and seven weeks at each study visit. Change will be evaluated between: (i) baseline, (ii) post-1 week, (iii) post washout crossover baseline, (iv) post 1 week, and (v) post 4 weeks.
  Subjects will be evaluated using clinical and laboratory safety testing at baseline and each subsequent study visit.
  Each participant will be tracked longitudinally during the study using clinical and laboratory safety parameters

SECONDARY OUTCOMES:
Polyamine levels in urine and blood | Baseline, one week, and one month
  Polyamine levels at each study visit
Serum lipidomics | baseline, one week, and one month
  targeted
CRP marker of inflammatory activity | Baseline, and one month
  C reactive protein
Evaluation of molecular biology and bioeffect signalling using untargeted and targeted Metabolomics | Baseline, one week, and one month. Change will be evaluated between: (i) baseline, (ii) post-1 week, (iii) post washout crossover baseline, (iv) post 1 week, and (v) post 4 weeks.
  Targeted analysis of spermidine, other polyamines, and approximately 250 other biomarkers using both mass spectrometry (MS) and nuclear magnetic resonance (NMR) spectroscopy detection technology.
  Untargeted analysis of small molecule biomarkers using MS detection.
  The metabolite profiles of each participant will be tracked longitudinally during the study and changes to targeted or untargeted metabolite profiles occurring between visits due to supplementation or washout from treatment will be evaluated.
Urinary untargeted and targeted metabolomics. Evaluation of molecular biology and bioeffect signalling and biomarker assessment | Baseline, one week, and one month. Change will be evaluated between: (i) baseline, (ii) post-1 week, (iii) post washout crossover baseline, (iv) post 1 week, and (v) post 4 weeks.
  Targeted analysis for small molecule biomarkers of human genomic, dietary and microbiome origin including amino acids (human), 2-furoylglycine (dietary), 3-hydroxyhippurate (microbial metabolism) and approximately 50 others using nuclear magnetic resonance (NMR) detection technology. Untargeted analysis of small molecule biomarkers of human genomic, dietary and microbiome origin using mass spectrometry (MS) and NMR spectroscopy detection.
Autophagy assay | Baseline and one week
  Western blot or Elisa assay

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kelley, MD, Principal Investigator — Biofortis Innovation Services Addison, IL, United States, 60101
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keohane P, Everett JR, Pereira R, Cook CM, Blonquist TM, Mah E. Supplementation of spermidine at 40 mg/day has minimal effects on circulating polyamines: An exploratory double-blind randomized controlled trial in older men. Nutr Res. 2024 Dec;132:1-14. doi: 10.1016/j.nutres.2024.09.012. Epub 2024 Sep 19. PMID 39405978